CLINICAL TRIAL: NCT03059563
Title: Dopamine D2/D3 Receptor Upregulation by Varenicline in Methamphetamine Users
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Global pandemic
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Edythe London, Professor of Psychiatry and Biobehavioral Sciences and Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-000445; 1R21DA042347-01A1 (NIH)
Record Dates: First submitted 2017-02-06; First posted 2017-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Dopamine D2/3 Receptor Availability; Cognitive Function; Methamphetamine Abuse
Keywords: Varenicline; Positron Emission Tomography; Functional Magnetic Resonance Imaging; Methamphetamine Abuse
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline (Experimental): A standard dose titration regimen that is used for smoking-cessation will be followed. The pharmacist will prepare capsules of varenicline for each week of study participation. Under observation by a study clinician, participants will receive one capsule containing 0.5 mg VAR each day (0900 h) for 3 days, then one capsule containing 0.5 mg VAR twice daily (0900 h, 2100 h) for 4 days, and finally a capsule containing 1 mg VAR twice daily (0900 h, 2100 h) for the next 2 weeks.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): The same procedure used for varenicline treatment will be followed. The pharmacist will prepare capsules of placebo for each week of study participation. Under observation by a study clinician, participants will receive one capsule containing placebo each day (0900 h) for 3 days, then one capsule containing placebo twice daily (0900 h, 2100 h) for 4 days, and finally a capsule containing placebo twice daily (0900 h, 2100 h) for the next 2 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline is an FDA-approved medication to facilitate smoking cessation. it is also a promising candidate to enhance dopamine signaling by upregulating dopamine D2/D3 (type 2) receptors in the striatum and improve cognitive function.
  Other Names: Chantix
  Arms: Varenicline
Other: Placebo — A placebo containing no active ingredients will be used as a control to assess the effects of varenicline on dopamine D2/D3 receptor availability and cognitive function.
  Arms: Placebo

SUMMARY:
While deficits in dopamine D2-type receptor availability have been linked to substance use disorders, higher availability associates with better behavioral treatment outcomes for stimulant dependence and resilience to addiction. Varenicline has been shown to upregulate D2-type receptors in drug-naive rats, and could be a useful therapeutic approach for the treatment of addictive disorders in humans.

The purpose of the study is to assess the relationship between varenicline, dopamine signaling (specifically, D2-type receptor availability), functional connectivity within corticostriatal circuitry, genetic markers associated with smoking and methamphetamine abuse, and measures of cognitive performance.

The investigators hypothesize that varenicline but not placebo will upregulate (increase) striatal dopamine D2-type receptor availability and improve cognition, and that the change in availability will correlate with the change in cognition. The investigators also hypothesize that varenicline but not placebo treatment will repair dysregulated connectivity between the striatum and prefrontal cortex observed in methamphetamine users, and will correlate with the change in cognition.

The study design consists of two positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) scans to measure dopamine D2-type receptor availability and functional connectivity between the prefrontal cortex and striatum, two cognitive testing sessions including a battery of tests assessing working memory, declarative memory, sustained attention, inhibitory control, and reward-based decision making. Following eligibility screening, thirty six methamphetamine users will be enrolled and tested/scanned once prior to initiation of varenicline or placebo treatment and then again after completion of treatment.

DETAILED DESCRIPTION:
1. Participants will be recruited from the Tarzana Treatment Center, the Domiciliary Residential Rehabilitation Program, or Chabad Treatment Center, where they will be residing in a residential substance use disorder program. Potential participants recently admitted with stimulant use disorder will be given a flyer describing the study, and interested parties will meet with a research associate to discuss details of the protocol and sign the informed consent form. Prior to enrollment, they will be screened for initial eligibility criteria and exclusion criteria. Participants who provide written consent will complete questionnaires about their mood, medical, psychiatric and drug use history, personality and life experiences. They will also give a urine sample to determine what drugs they have recently used, a breath sample to determine the carbon monoxide levels in their system, and a blood sample to assess complete blood count, metabolic panel, screening for infectious diseases, and tests of kidney function. This blood sample will also be used to determine follicular and luteal phase in female participants.
2. Consenting participants will meet with the study physician for additional screening. The study physician will take a medical history, take a personal and family health profile, perform a physical examination, and collect and review laboratory tests to determine eligibility.
3. Participants will be seen at least weekly for follow-up throughout the study via a set of self-report questionnaires, including the Mini International Neuropsychiatric Interview (MINI), Patient Health Questionnaire-9, 4-Item Positive Symptom Rating Scale, Mood Disorder Questionnaire, International Physical Activity Questionnaire, and side effect questionnaires. Urine samples and exhaled breath will also be collected at these follow-up visits.
4. After completing screening procedures, eligible participants will complete the following baseline assessments:

   A) Visit 1:

   i. Structural magnetic resonance imaging (MRI): High-resolution structural MRI scans of the brain Magnetization-Prepared Rapid Acquisition Gradient Echo will be obtained before positron emission tomography (PET) scans to confirm the absence of structural brain lesions and to aid in localization of volumes of interest.

   ii. Functional MRI (fMRI): The purpose of this session is to collect information on brain function and activity while participants are engaged in cognitive tasks and at rest, while accounting for physiological variability. During the scan, non-invasive physiological measurements, including respiration, pulse and rate of eye blinks will be collected to determine signals in fMRI data related to physiology. Resting state scans will be acquired to examine the functional connectivity of brains regions in the absence of cognitive demands. Participants will be asked to stare at a black screen. Participants will be asked to smoke 15-30 minutes prior to the fMRI scan.

   Participants may be asked to complete two or three of the following cognitive tasks in the scanning environment:

   The Balloon Analog Risk Task (BART): The BART measures risky decision making. During the BART, participants must make a series of choices between two options: inflating a virtual balloon to increase potential monetary gains ($0.25/inflation) or not inflating a virtual balloon and retaining accrued earnings. Each time a virtual balloon is inflated, the size and value of the balloon increases or the balloon explodes and the participants earn no money on that trial. The task will be administered in one 10-minute session.

   Reversal Learning task (RLT): Participants perform a simple categorization task with reversal stages. Participants learn to make one of two key-press responses to a set of abstract visual patterns (e.g., fractal patterns) on the basis of trial-by-trial feedback. Subjects view the stimuli (which are novel visual patterns) and must make a key press. Immediately after the response, feedback will appear on the screen: "correct", "incorrect", or a "no response recorded" message if no response is made within the response window. Participants will be trained on these stimuli that have varying numbers of trials before the reversal phase. The reversal phase is unbeknownst to the participant where previously correct stimuli are now incorrect. Participants learn this new pattern through feedback. After the task, participants may participate in a memory test of the pictures they saw during the RLT.

   Stop Signal Task (SST): This task consists of 256 trials (64 Stop trials). Each trial will begin with a fixation dot appearing at the center of the screen for 500 milliseconds (ms), followed by a target stimulus, "O" or "X", which will remain for 2000ms. Participants will be instructed to respond as quickly as possible with a left key-press for "O" or a right key-press for "X", but to try to stop themselves from pressing if the target was followed by a "stop-signal" tone (25% of trials). This signal will be presented at a variable delay (the stop-signal delay), after the target stimulus appears. After a successful Stop trial, the stop-signal delay will be increased by 50ms, and after a failed Stop trial, it will be decreased by 50ms, eventually titrating to a stop-signal delay resulting in ~50% successful inhibition rate. 3 days prior to the fMRI visit, each participant will be trained on this task.

   B) Visit 2:

   i. Prior to completing behavioral tasks and PET scanning, participants will visit the Clinical and Translational Research Center, where a registered nurse will draw approximately 20 milliliters (mL) of blood. Blood samples will be tested for plasma levels of nicotine, cotinine, and trans-3'-hydroxycotinine, as well as genetic markers associated with smoking and methamphetamine use.

   The DNA samples acquired from this protocol will be added to a larger database of DNA samples collected from participants in London Laboratory protocols. DNA samples will be stored for future use other than the aims and goals of this study. Participants will not receive their results because our laboratory is only qualified for genetic analyses associated with research purposes and is not certified for clinical assessment of genetic information.

   This blood sample will also be used to determine follicular and luteal phase in female participants.

   ii. Cognitive/behavioral testing: Working memory (N-back test), declarative memory (Rey Auditory Verbal Learning Task),sustained attention (Rapid Visual Information Processing), inhibitory control (Stop Signal Test) and reward-based decision-making (Monetary Delay Discounting and Reversal Learning) will be tested on the same day of the PET scan.

   iii. PET Scanning: A computed tomography transmission scan will be performed, before administration of the radiopharmaceutical, to obtain data for measured attenuation correction. A dose of [18F]fallypride, approximately 5 millicuries (mCi) (+/- 10% error) with an injected mass of 1.82 micrograms (μg) (+/- 10% error), will be administered as an intravenous bolus injection. Dynamic scanning will start after the bolus injection. The first dynamic emission scanning sequence will take 80 min. The participant will then be removed from the scanner for a 20-minute break. To reduce radiation-absorbed dose to the urinary bladder wall, participants will be instructed to water load and void during their break. A second 80-minute dynamic emission scan acquisition will follow.
5. Participants will be randomly assigned to a varenicline (VAR) treatment or placebo group by the Semel Institute Statistic Unit. The participant as well as the experimenters administering PET scans or cognitive tests will be blinded to the assigned treatment. Both conditions will require that participants take capsules as instructed over the course of 3 weeks. Medications (active and placebo) for the upcoming week will be dispensed at the beginning of each week. At the end of each week, the participants will meet with the study physician for a check-up to monitor potential adverse events. After the 3-wk regimen (VAR or placebo), participants will undergo repeat testing of PET measures and behavioral tests as described in section 6. On the final day of treatment, a blood sample will be taken to assess plasma levels of VAR.
6. After completing VAR treatment, participants will complete the following assessments:

   A) Visit 3:

   i. Structural MRI. As described in Visit 1.

   ii. Functional MRI (fMRI): As described in Visit 1.

   B) Visit 4:

   i. Prior to completing behavioral tasks and before undergoing PET scanning, participants will visit the Clinical and Translational Research Center, where a registered nurse will draw approximately 20 mL of blood. Blood samples will be sent to the Tyndale laboratory and tested for plasma levels of varenicline, and plasma levels of nicotine, cotinine, and trans-3'-hydroxycotinine to assess changes in smoking status from baseline. This blood sample will also be used to determine follicular and luteal phase in female participants.

   ii. Cognitive/behavioral testing As described in Visit 2.

   iii. PET Scanning: As described in Visit 2.
7. Participants will be reimbursed for transportation costs to the University of California, Los Angeles from their inpatient treatment center throughout the entirety of the study. They will be escorted with a research associate via a taxi cab.

ELIGIBILITY:
Inclusion Criteria:

* English fluency in order to provide informed consent and complete questionnaires
* Age of 18-60 years [Children younger than 18 years will be excluded because of the potential risk of radiation exposure. Recruitment will be restricted to individuals within the first 5 decades of life to avoid effects of aging on DRD2/3 (dopamine type-2 receptor) BPND (binding potential).
* Meeting DSM (Diagnostic and Statistical Manual of Mental Disorders) 5 criteria for stimulant-use disorder
* Being within 2 weeks of admission to treatment and < 2 months abstinent from stimulant use
* Vital signs as follows: resting pulse between 50 and 95 beats per minute (bpm), blood pressures between 90-150 mm Hg (millimeter of mercury) systolic and 45-95 mm Hg diastolic
* Hematology and chemistry laboratory test results within normal (+/- 10%) limits and normal kidney function (estimated glomerular filtration rate ≥ 90 ml/min/1.73m2)
* Baseline ECG (electrocardiogram) demonstrating normal conduction (including QTc [QT interval]) without clinically significant arrhythmias
* Absence of clinically significant contraindications for participation, in the judgment of the admitting physician and the principal investigator, assessed by a medical history and physical examination.

Exclusion Criteria:

* History or evidence of seizure disorder or brain injury with loss of consciousness >30 min
* Previous adverse reaction to varenicline (VAR)
* Neurological disorder that would compromise informed consent or complicate data interpretation (e.g., organic brain disease or dementia)
* Past-year psychotic disorder assessed by the Mini-International Neuropsychiatric Interview (MINI)
* History of a suicide attempt and/or current suicidal ideation or plan, as assessed by the MINI
* Evidence of clinically significant heart disease or hypertension, as determined by physical exam, or ECG showing cardiac ischemia or other clinically significant abnormality, or use of warfarin
* Evidence of untreated or unstable medical illness, including endocrine, autoimmune, renal, hepatic, or active infectious disease which might compromise safety during participation, as determined by history and physical examination and laboratory tests
* Diabetes or use of insulin
* Pregnancy or nursing [Note: Female participants must be either postmenopausal or using a reliable form of contraception (e.g., abstinence, oral contraceptive pills, intrauterine device, sterilization, condoms or spermicide). Women must have negative urine tests for pregnancy at study entry and on positron emission tomography (PET) scan days]
* Asthma or use of theophylline, α- or β-adrenergic agonists, or other sympathomimetics; 12) use of any medications (e.g., neuroleptics) that directly affect dopaminergic neurotransmission in brain; 13) claustrophobia [Participants will be questioned about their potential discomfort if in an enclosed space, such as a PET or magnetic resonance imaging (MRI) scanner]
* Exceed radiation exposure limits [Participation in any other research involving exposure to ionizing radiation in the past year will be exclusionary if the total cumulative exposure from the past and current research would exceed the limits set by the Food and Drug Administration in 21 Code of Federal Regulations 361.1. The total cumulative dose to the whole body, active blood-forming organs, lens of the eye, and gonads must remain < 5 rems, and the cumulative dose to all other organs must remain < 15 rems. Volunteers who were exposed to ionizing radiation in the year before potential entry to this study will be excluded if they cannot provide proper documentation of the amount of past research radiation exposure.]
* A metal device (e.g., pacemaker, infusion pump, aneurysm clip, prosthesis or plate) in the body [Presence of such a device could either interfere with scan acquisition or pose a potential risk during MRI. A participant who has an implanted device can enroll if s/he provides documentation that the device is MRI-compatible.];
* Any condition that, as deemed by the investigators and study physician, would compromise safe participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Dopamine D2-type receptor availability | 21 days
  Dopamine D2-type receptor binding potential in the striatum measured with positron emission tomography scanning measured at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.

SECONDARY OUTCOMES:
Sustained attention | 21 days
  The Continuous Performance Task will be used to assess sustained attention at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Working memory | 21 days
  The Sternberg Spatial task will be used to assess working memory at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Declarative memory | 21 days
  The Rey Auditory Verbal Learning Test will be used to assess declarative memory at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Inhibitory control - stop signal task | 21 days
  The Stop-signal task will be used to assess inhibitory control at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Inhibitory control - reversal learning | 21 days
  A reversal learning task will be used to assess inhibitory control at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Reward-based decision-making | 21 days
  A monetary delay-discounting task and the Balloon Analogue Risk task will be used to assess reward-based decision-making at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Resting state functional connectivity | 21 days
  Striatum resting state functional connectivity will be measured with a functional magnetic resonance imaging scan at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Task-based brain activity (functional magnetic resonance imaging) - balloon analog risk | 21 days
  Performance on a cognitive task (the Balloon Analog Risk Task) will be assessed during a functional magnetic resonance imaging scan at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Task-based brain activity (functional magnetic resonance imaging - stop signal | 21 days
  Performance on a cognitive task the (Stop Signal Task), will be assessed during a functional magnetic resonance imaging scan at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Decision making under risk and ambiguity | 21 days
  A task involving decision making under during differing types of risk and ambiguity will be used to determine decision making under risk and ambiguity at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.
Loss Aversion | 21 days
  A computer task and written questionnaire assessing loss preferences will be used to assess loss aversion at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment.

OTHER OUTCOMES:
Personality - impulsivity | 21 days
  Self-report of impulsivity will be measured at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment using the Barratt Impulsiveness Scale.
Personality - novelty seeking | 21 days
  Self-report of novelty seeking will be measured at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment using the Temperament and Character Inventory.
Personality - reward dependence | 21 days
  Self-report of reward dependence will be measured at baseline prior to varenicline/placebo and after 3 weeks of varenicline/placebo treatment using the Temperament and Character Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States